CLINICAL TRIAL: NCT03902470
Title: Comparative Study Between Awake Thoracic Epidural Anaesthesia and General Anesthesia for Video Assisted Thoracoscopic Surgery
Brief Title: Awake Thoracic Epidural Anaesthesia Versus General Anesthesia for Video Assisted Thoracoscopic Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, rabeea ahmed Mohamed, Resident at assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anesthesia for VATS
Record Dates: First submitted 2019-03-21; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: In determining a significant difference (20%) in the occurrence of postoperative pain score by using the power of 80% and a significance level of 5% and this will result in 30 patients in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural anaesthesia for vats (Experimental): Patients in thoracic epidural (TE) group will pre-medicated using midazolam 3-4 mg intravenous (IV)and fentanyl 50 mcg intravenously(i.v.). Then patients will placed in the lateral decubitus position. An epidural catheter will be inserted between T3-T4 and T4-T5 for all thoracic procedures except sympathectomy and thymectomy. A test dose (5 ml) of 2% lidocaine will be given, followed by 15-20 ml of bupivacain 0.5% and 50 mcg of fentanyl.
  The objective is to achieve sensory and motor block between C7 and T7 levels. At this level diaphragmatic respiration is maintained. The anaesthesia level will be monitored by warm-cold discrimination.
  Interventions: Procedure: Thoracic epidural anaesthesia video assisted thoracoscopic surgery
- General anesthesia for vats (Active Comparator): Patients will receive general anesthesia as follows, Premedication in the form of 3-4 mg midazolam (IV), induction of a anesthesia with propofol (2mg/kg) and fentanyl (1 mcg/kg). Tracheal intubation and double endotracheal tube insertion will be facilitated with cisatracurium 0.1 mg/kg. and confirmation of it is position will made by fiberoptic bronchoscopy, Anesthesia will be maintained with isoflurane (1-2 %) and cisatracurium (0.05 mg/kg per dose).After the end of the operation, anesthesia will be discontinued, the wound dressing will be applied, and extubation of the patient will be done after reversal of muscle relaxant by neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg) and extubation will be performed after complete neuromuscular recovery.
  Interventions: Procedure: Thoracic epidural anaesthesia video assisted thoracoscopic surgery

INTERVENTIONS:
Procedure: Thoracic epidural anaesthesia video assisted thoracoscopic surgery — Patients in (TEA) group will pre-medicated using midazolam 3-4 mg (IV)and fentanyl 50 mcg (IV). Then An epidural catheter will be inserted between T3-T4 and T4-T5 . A test dose (5 ml) of 2% lidocaine will be given, followed by 15-20 ml of bupivacain 0.5%.

SUMMARY:
Thoracic procedures are routinely performed under general anesthesia (GA), with one lung ventilation (OLV)by double lumen tube or (GA) in spontaneously breathing patient by TIVA or LMA are usually combined with thoracic epidural analgesia.

However, GA whether mechanically ventilated or spontaneously breathing may have adverse effects including peri-intubation hypoxia, trauma to the upper airway, mechanical ventilation-induced injuries, impaired cardiac performance, neuromuscular problems in OLV and increased risk of pneumonia, and release of proinflammatory mediators in generally.

Recently, awake thoracic epidural anesthesia (ATEA) has been used alone in thoracic procedures The results achieved in early studies have been encouraging. ATEA may eventually provide an alternative method to GA for thoracic procedures that would not only eliminate the need for GA but also facilitate both surgical reconstruction and eventually patient recovery.

Recent studies suggested better clinical outcomes with ATEA, including less intraoperative bleeding, a better control of postoperative pain, early mobilization and short hospital stay, oral intake tolerance, reduction of surgical stress response, reduction of intraoperative cardiac events, improvement of myocardial flow determinants and left ventricular function, and a reduction of complications including pulmonary, thrombotic and infectious events.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 60 years.
* ASA score equal to or less than III.
* The absence of severe emphysema or clinical signs of active infectious disease.
* The procedure is predicted to be completed within two hours.

Exclusion Criteria:

* Patients with expected difficult airway management
* Haemodynamically unstable patients
* Obesity (body mass index >30)
* Inexperienced and poorly cooperative surgical team
* Coagulopathy (international normalized ratio >1.5)
* Persistent cough or high airway secretion
* Neurological disorders: risk of seizure, unable to cooperate, intracranial mass or brain oedema
* Extensive pleural adhesions or previous pulmonary resections
* Hypoxaemia (PaO2 <60) or hypercarbia (PCO2 >50)
* Any contraindications for use of regional anesthesia technique

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Recovery time after intervention of each group | 7days
  The time of anesthesia recovery, resumption of oral intake,and the length of hospital stay,postoperative recovery index will be used will be used to assess recovery as next Higher scores reflect greater difficulty in post-operative recovery
  No Difficulty 1 Little Difficulty >1 to <1.5 Moderate Difficulty 1.5 to <2.5 Considerable Difficulty 2.5 to <3.5 Extreme Difficulty 3.5 to 5 PoRI Scale and Subscale Scoring System.

SECONDARY OUTCOMES:
Patient agitation and sedation by using richmond agitation-sedation scale(RASS) | 4 hourly postoperative.
  1. Observe patient
  1. Patient is alert, restless, or agitated. (Score 0 to +4) 2. If not alert, state patient's name and say to open eyes and look at speaker.
  2. Patient awakens with sustained eye opening and eye contact. (Score -1)
  3. Patient awakens with eye opening and eye contact, but not sustained. (Score -2)
  4. Patient has any movement in response to voice but no eye contact. (Score -3) 3. When no response to verbal stimulation, physically stimulate patient by shaking shoulder and/or rubbing sternum.
  5. Patient has any movement to physical stimulation. (Score -4)
  6. Patient has no response to any stimulation. (Score -5)

OTHER OUTCOMES:
Incidence of complications | 14days
  Impaired cardiac performance assessed by Echo and incidence of pneumonia assessed by chest x-ray.

IPD SHARING:
Plan to Share IPD: Undecided